CLINICAL TRIAL: NCT04014673
Title: Natural History Characterization in Symptomatic and Asymptomatic Progranuline Gene Mutation Carriers
Acronym: Predict-PGRN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P071229
Record Dates: First submitted 2019-04-15; First posted 2019-07-10 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Frontotemporal Lobar Degeneration
Keywords: Frontotemporal Dementia,; biomarkers,; brain Imaging PET
MeSH Terms: conditions — Frontotemporal Lobar Degeneration; Frontotemporal Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with a PGRN gene mutation (Other): Symptomatic patients with a PGRN gene mutation
  Interventions: Behavioral: Behavioral : Characterization
- Presymptomatic individuals (Other): Asymptomatic 'At-risk' individuals with a PGRN gene mutation
  Interventions: Behavioral: Behavioral : Characterization
- healthy volunteers (Other): 'At-risk' individuals without a PGRN gene mutation
  Interventions: Behavioral: Behavioral : Characterization

INTERVENTIONS:
Behavioral: Behavioral : Characterization — Behavioral scales and neuropsychological tests; MRI, SPECT/PET

SUMMARY:
The purpose of this study is to investigate whether cognitive deficits, structural and functional changes can be detected before symptom onset in presymptomatic progranuline mutation carriers. The main objectives of the project are to identify novel cognitive, brain imaging markers and peripheral biomarkers for early diagnosis of FTLD, and to follow disease progression.

DETAILED DESCRIPTION:
The project focuses on the progranulin (PGRN) gene mutation, one of the most frequent genetic forms of frontotemporal dementias (FTD, or frontotemporal lobar degeneration, FTLD). FTD is the second commonest cause of degenerative dementia in presenium after Alzheimer's disease. Behavioral and cognitive impairments progressively lead to dementia. Two major pathological subtypes are now defined in FTD, FTD-TDP and FTD-TAU.

FTD is difficult to detect at an early stage, and no clinical, biological or imaging features can predict the underlying pathology in living patients. Therapeutic perspectives have emerged against tau aggregation, PGRN deficit and C9orf72 expansion. Presymptomatic carriers of genetic FTD would benefit, before onset of symptoms, from these therapeutics that would delay or prevent the disease. At this step, it becomes crucial to develop markers to know how many years before symptoms, the pathological process begins, to treat the patients at the earliest stage of the disease. Markers are also needed to predict the pathology (FTD-TDP/FTD-tau) in patients that will be eligible for trials targeting specific pathological lesion. The main objectives of the project are to identify novel cognitive, brain imaging markers and peripheral biomarkers for early diagnosis of FTLD, and to follow disease progression. Ninety participants including 8 patients and 82 'at-risk' individuals will be recruited and evaluated by clinical partners of the project (Paris, Lille, Rouen, Toulouse, Saint-Etienne, Marseille, Nantes). 'At-risk individuals' are the first- degree relatives of PGRN patients, who have a high a risk (50%) to carry the mutation.

Brain structural changes will be evaluated by voxel-based morphometry (SPM12 software) to assess global brain atrophy in one with the evaluation of atypical shape patterns such as cortical thickness (Freesurfer software) and the study of the cortical sulci (BrainVISA/Morphologist software).

Fluoro Deoxy DGlucose-Positron Emission Tomography (FDG-PET) will allow the identification of brain metabolic markers. Then voxel-based methods using Statistical Parametric Mapping software will be applied to compare different groups or analyze correlations between brain metabolism and cognitive deficits.

The identification of peripheral biomarkers of disease onset and disease progression will take advantage from RNA sequencing, in order to study gene expression and RNA splicing alterations in lymphocytes of patients and 'at risk individuals'.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for symptomatic patients:

* Age ≥ 18
* Signed informed consent for genetic and clinical study
* To be carrier of a PGRN mutation - Diagnosis criteria of FTD
* To be affiliated to the social security scheme

Inclusion criteria for 'at-risk' asymptomatic relatives:

* Age ≥ 18
* To be first degree relative of a person carrying a PGRN mutation or first degree relative of FTD deceased patient whose PGRN mutation as been identified in the family
* Signed informed consent for genetic and clinical study
* To be affiliated to the social security scheme

Exclusion Criteria:

Exclusion criteria for symptomatic patients:

* Presence of one exclusion criteria from Diagnosis criteria of FTD. - Participation to another therapeutic trial. - Contra-indication to perform a brain MRI and/or PET-FDG
* Inability to lie one hour without moving
* Breastfeeding and pregnant women
* Presence of another intercurrent neurological pathology (vascular cerebral accident, tumor, etc.....)

Exclusion criteria for 'at-risk' asymptomatic relatives :

* Presence of neurological or neurodegenerative disease
* Clinical proven signs of FTD, language disorder, praxis disorder, mnemic, of parkinson's syndrome or amyotrophic lateral sclerosis
* Contra-indication to perform a brain MRI and/or PET-FDG
* Inability to lie one hour without moving
* Breastfeeding and pregnant women
* Severe vascular lesion , tumor or infectious brain imaging if an MRI was done previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-01-19 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Rate of change of Frontal Assessment Battery score (/18) | at baseline 0 Months,at 42 Months,at 72 Months
  Executive functions changes over time (rate of change in neuropsychological test)
Rate of change of Trail Making Test B-A time (seconds) | at baseline 0 Months,at 42 Months,at 72 Months
  Cognitive flexibility changes over time (rate of change in neuropsychological test)
Rate of change of Ekman's faces test score (/35) | at baseline 0 Months,at 42 Months,at 72 Months
  Emotional assessment changes over time (rate of change in neuropsychological test)
Rate of change of Faux-pas test score (/35) | at baseline 0 Months,at 42 Months,at 72 Months
  Social cognition changes over time (rate of change in neuropsychological test)
Rate of change of Digit span score | at baseline 0 Months,at 42 Months,at 72 Months
  Short-term memory changes over time (rate of change in neuropsychological test)
Rate of change of Free and Cued Selective Reminding test, total recall score (/48) | at baseline 0 Months,at 42 Months,at 72 Months
  Long-term memory changes over time (rate of change in neuropsychological test)
Rate of change of Boston Naming test score (/34) | at baseline 0 Months,at 42 Months,at 72 Months
  Language changes over time (rate of change in neuropsychological test)
Rate of change of Gestural Praxis battery score (/168) | at baseline 0 Months,at 42 Months, at 72 Months
  Gestural praxis changes over time (rate of change in neuropsychological test)
Rate of change of Neuropsychiatric Inventory score (/144) | at baseline 0 Months,at 42 Months,at 72 Months
  Behavioral changes over time (rate of change in neuropsychological questionnaire)
Rate of change of Apathy Evaluation Scale score (/42) | at baseline 0 Months,at 42 Months,at 72 Months
  Apathy changes over time (rate of change in neuropsychological questionnaire)
Change in MRI morphological criteria (brain atrophy by voxel-based morphometry) | at baseline 0 Months,at 42 Months,at 72 Months
Change in cerebral metabolism by PET (metabolic markers by Fluoro-DeoxyDGlucose-Positron Emission Tomography (FDG-PET)) | at baseline 0 Months,at 42 Months,at 72 Months

SECONDARY OUTCOMES:
Correlations between cognitive and behavioral scores, MRI morphological criteria, cerebral metabolism by FDG-PET and transcriptome analysis in presymptomatic subjects and in symptomatic patients at early disease stage | at baseline 0 Months,at 42 Months,at 72 Months
  Voxel-based methods using Statistical Parametric Mapping software will be applied to compare different groups or analyze correlations between brain atrophy/metabolism and cognitive deficits.
Differences in transcriptome analysis between symptomatic patients, asymptomatic carriers and controls. | at baseline 0 Months,at 42 Months,at 72 Months
  Study gene expression and RNA splicing alterations in lymphocytes (RNA sequencing)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle LE BER, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Groupe Hospitalier Pitié-Salpêtrière - Charles Foix, Paris
  - Pitié Salpetriere Hospital, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caroppo P, Habert MO, Durrleman S, Funkiewiez A, Perlbarg V, Hahn V, Bertin H, Gaubert M, Routier A, Hannequin D, Deramecourt V, Pasquier F, Rivaud-Pechoux S, Vercelletto M, Edouart G, Valabregue R, Lejeune P, Didic M, Corvol JC, Benali H, Lehericy S, Dubois B, Colliot O, Brice A, Le Ber I; Predict-PGRN study group. Lateral Temporal Lobe: An Early Imaging Marker of the Presymptomatic GRN Disease? J Alzheimers Dis. 2015;47(3):751-9. doi: 10.3233/JAD-150270. PMID 26401709
- [Result] Saracino D, Sellami L, Boniface H, Houot M, Pelegrini-Issac M, Funkiewiez A, Rinaldi D, Locatelli M, Azuar C, Causse-Lemercier V, Jaillard A, Pasquier F, Chastan M, Wallon D, Hitzel A, Pariente J, Pallardy A, Boutoleau-Bretonniere C, Guedj E, Didic M, Migliaccio R, Kas A, Habert MO, Le Ber I; Predict-PGRN. Brain Metabolic Profile in Presymptomatic GRN Carriers Throughout a 5-Year Follow-up. Neurology. 2023 Jan 24;100(4):e396-e407. doi: 10.1212/WNL.0000000000201439. Epub 2022 Oct 18. PMID 36257714
- [Derived] Saracino D, Dorgham K, Camuzat A, Rinaldi D, Rametti-Lacroux A, Houot M, Clot F, Martin-Hardy P, Jornea L, Azuar C, Migliaccio R, Pasquier F, Couratier P, Auriacombe S, Sauvee M, Boutoleau-Bretonniere C, Pariente J, Didic M, Hannequin D, Wallon D; French Research Network on FTD/FTD-ALS; PREV-DEMALS and Predict-PGRN study groups; Colliot O, Dubois B, Brice A, Levy R, Forlani S, Le Ber I. Plasma NfL levels and longitudinal change rates in C9orf72 and GRN-associated diseases: from tailored references to clinical applications. J Neurol Neurosurg Psychiatry. 2021 Dec;92(12):1278-1288. doi: 10.1136/jnnp-2021-326914. Epub 2021 Aug 4. PMID 34349004